CLINICAL TRIAL: NCT06511557
Title: Comparative Effect of Non Immersive Virtual Reality Based Training (Xbox Kinect) and Kinetic Chain Exercises in Patient With Knee Osteoarthritis.
Brief Title: Comparison of Effect of Virtual Reality and Kinetic Chain Exercises in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS /23/01115
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Xbox kinetic; Virtual Reality Rehabilitation; Kinetic chain exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Clinical study in which two or more groups of participants receive different interventions. Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial. Assignment to a group usually is randomized
Who Masked: Outcomes Assessor
Masking Description: Masking refers to a practice where study participants are prevented from knowing certain information that may somehow influence them thereby tainting the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non immersive virtual reality (Xbox kinetic) (Experimental): * Track and field.
  * Skiing.
  * Dance Central.
  * Kinect sports.
  Interventions: Device: Non immersive virtual reality ( xbox kinetic)
- Kinetic Chain Exercises (Active Comparator): Closed chain:
  Terminal Knee Extension.
  * Semi squat.
  * Forward step up and down.
  Open chain:
  * SLR in lying.
  * Knee extension in sitting.
  Interventions: Other: Kinetic chain exercises

INTERVENTIONS:
Device: Non immersive virtual reality ( xbox kinetic) — Treatment starts with a gentle warm-up i.e. hot pack for 10 minutes and gentle stretching of Quadriceps, hamstrings and calves. Each game was performed for 10 minutes with 1 minute rest between games. 3 sessions Per Weeks for 8 weeks (45 Min per Session) were given. All the exergames target muscles like Hamstring, Quadriceps and calves to improve function of knee joint and reduce pain.
  Baseline assessment was done at the start of the session and proper cool down and stretching will be performed at the end of each session to promote flexibility and reduce muscle soreness
  Arms: Non immersive virtual reality (Xbox kinetic)
Other: Kinetic chain exercises — Session starts with a gentle warm-up i.e. Hot pack for 10 minutes and gentle stretching. Each exercise is performed in 2 sets, each set of 10 repetitions with 1min rest between sets. 3 sessions Per Weeks for 8 weeks (45 Min Per Session) were given .Kinetic chain exercises involve integrated movements that engage multiple joints and muscle groups & focus on strengthening muscles like quadriceps, hamstrings, glutes, and calf muscles, improving joint stability, function, and reducing pain. Baseline assessment was done at the start of the session and proper cool down and stretching was performed at the end of each session to promote flexibility and reduce muscle soreness
  Arms: Kinetic Chain Exercises

SUMMARY:
It is necessary to explore the novel rehabilitation strategies to treat knee osteoarthritis. Although kinetic chain exercises have shown efficacy but there is growing interest in Virtual Reality training using Xbox Kinect because it has the potential to enhance motivation and patient's adherence to Rehabilitation. The aim of this study is to compare the effectiveness of both interventions and provide a valuable insight to optimize the therapeutic strategies for treating knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a prevalent musculoskeletal condition that impacts the quality of life. Despite various treatment options, managing knee OA is still a challenge for healthcare professionals. However, there is growing interest in exploring the innovative interventions to decrease symptoms and improve functional outcome in patients with knee OA.The project will be a Randomized control trial conducted to check the effect of Virtual Reality and Kinetic chain exercises in patients with knee osteoarthritis.so that we can have best treatment option. Duration of this study will be of 8 weeks , convenient sampling will be done, subjects following eligibility criteria from IIMCT Pakistan Railway general Hospital will be randomly allocated in two groups, baseline assessment will be done, Group A will be given Xbox kinetic training and Group B will be given Kinetic chain exercises . Outcome measures if this research will be pain , Range if Motion , function and disability. Post intervention assessment will be done via NPRS , WOMAC , KOOS_PS and goniometric measurements of Knee ranges .Data was analyzed by using SPSS software. There is lack of research comparing the effectiveness of Virtual Reality Xbox Kinect and kinetic chain exercises in patients with knee osteoarthritis. There are studies that have explored the effectiveness of these interventions separately. In past, few researches support the fact that virtual reality rehabilitation is more effective than conventional physical therapy and few researches are in support of kinetic chain exercises being more effective for knee osteoarthritis. However there is no study that has compared these both interventions. Therefore there is a need for further research to compare both of these interventions which in future will provide optimal, more personalized and effective rehabilitation strategy for individuals with knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Both male & female

  * Age 50 or older.
  * Body mass index (BMI) between 18.9kg/m2 and 29.9 kg/m2.
  * Diagnosed with Grade II knee OA
  * Have knee pain > 4 on NPRS
  * Ability to engage in moderate physical activity.

Exclusion Criteria:

* Severe comorbidities limiting physical activity.

  * History of Hip and Knee arthroplasty.
  * Cognitive impairments affecting comprehension

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale: | [Time Frame: 8 weeks]
  The Numeric Pain Rating Scale (NPRS) is used to assess pain. On an 11-point Numeric scale, 0 represents no pain and 10 Represents the worst imaginable pain.
Knee injury and Osteoarthritis Outcome score (KOOS PS): | [Time Frame: 8 weeks]
  It is a self- administered questionnaire, designed for the assessment of individuals with knee osteoarthritis and injury. It consists of five subscales such as Pain, Activities of daily living , Symptoms, Sport and recreational activities and Quality of life related to knee. The KOOS short form typically consists of 7 questions covering five domains:
  Pain: 1 question Other Symptoms: 1 question Function in Daily Living (ADL): 1 question Function in Sport and Recreation (Sport/Rec): 2 questions Knee-related Quality of Life (QOL): 2 questions Each question is scored on a Likert scale ranging from 0 to 4, with 0 indicating no symptoms and 4 indicating extreme symptoms. The total score for the KOOS short form can range from 0 to 28 but we use reverse percentage for scoring which is from 0 to 100 precent with higher scores indicating greater severity in knee function.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): | [Time Frame: 8 weeks]
  It is a self-administered questionnaire widely used for the assessment of Health status of individuals With Osteoarthritis of Hip or Knee. It has three subscales such as Pain, Stiffness and Physical Function.
  The WOMAC questionnaire consists of 24 questions divided into three subscales:
  Pain (5 questions) Stiffness (2 questions) Physical Function (17 questions) Each question is answered on a Likert scale ranging from 0 to 4, with 0 indicating no symptoms and 4 indicating extreme symptoms. Therefore, the total score for the WOMAC index can range from 0 to 96, with higher scores indicating greater severity of osteoarthritis symptoms.
Range of Motion (Goniometer): | [Time Frame: 8 weeks]
  It is employed as a benchmark technique for the assessment of Range of motion of a joint, measured using a goniometer. Goniometer measures the joint ranges in every plane of the joint , it's measurements are highly reliable.

CONTACTS AND LOCATIONS:
Overall Officials: syed shakil urrehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- IIMCT Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim WB, Al-Dadah O. Conservative treatment of knee osteoarthritis: A review of the literature. World J Orthop. 2022 Mar 18;13(3):212-229. doi: 10.5312/wjo.v13.i3.212. eCollection 2022 Mar 18. PMID 35317254
- [Background] Hall M, van der Esch M, Hinman RS, Peat G, de Zwart A, Quicke JG, Runhaar J, Knoop J, van der Leeden M, de Rooij M, Meulenbelt I, Vliet Vlieland T, Lems WF, Holden MA, Foster NE, Bennell KL. How does hip osteoarthritis differ from knee osteoarthritis? Osteoarthritis Cartilage. 2022 Jan;30(1):32-41. doi: 10.1016/j.joca.2021.09.010. Epub 2021 Sep 29. PMID 34600121
- [Background] Ozudogru A, Gelecek N. Effects of closed and open kinetic chain exercises on pain, muscle strength, function, and quality of life in patients with knee osteoarthritis. Rev Assoc Med Bras (1992). 2023 Jul 17;69(7):e20230164. doi: 10.1590/1806-9282.20230164. eCollection 2023. PMID 37466598
- [Background] Ng WH, Jamaludin NI, Sahabuddin FNA, Ab Rahman S, Ahmed Shokri A, Shaharudin S. Comparison of the open kinetic chain and closed kinetic chain strengthening exercises on pain perception and lower limb biomechanics of patients with mild knee osteoarthritis: a randomized controlled trial protocol. Trials. 2022 Apr 15;23(1):315. doi: 10.1186/s13063-022-06153-8. PMID 35428274
- [Background] Byra J, Czernicki K. The Effectiveness of Virtual Reality Rehabilitation in Patients with Knee and Hip Osteoarthritis. J Clin Med. 2020 Aug 14;9(8):2639. doi: 10.3390/jcm9082639. PMID 32823832
- [Background] Raposo F, Ramos M, Lucia Cruz A. Effects of exercise on knee osteoarthritis: A systematic review. Musculoskeletal Care. 2021 Dec;19(4):399-435. doi: 10.1002/msc.1538. Epub 2021 Mar 5. PMID 33666347
- [Background] van den Bosch MHJ. Osteoarthritis year in review 2020: biology. Osteoarthritis Cartilage. 2021 Feb;29(2):143-150. doi: 10.1016/j.joca.2020.10.006. Epub 2020 Nov 24. PMID 33242602
- [Background] Dantas LO, Salvini TF, McAlindon TE. Knee osteoarthritis: key treatments and implications for physical therapy. Braz J Phys Ther. 2021 Mar-Apr;25(2):135-146. doi: 10.1016/j.bjpt.2020.08.004. Epub 2020 Sep 8. PMID 33262080
- [Background] Nambi G, Abdelbasset WK, Elsayed SH, Khalil MA, Alrawaili SM, Alsubaie SF. Comparative effects of virtual reality training and sensory motor training on bone morphogenic proteins and inflammatory biomarkers in post-traumatic osteoarthritis. Sci Rep. 2020 Sep 28;10(1):15864. doi: 10.1038/s41598-020-72587-2. PMID 32985509